CLINICAL TRIAL: NCT04275635
Title: Validation of a Predictive Algorithm to Determine the Effectiveness of Orthokeratology for Myopia Control
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Clinical investigator, Sun Yat-sen University
Other Study IDs: 2020KYPJ018
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children with myopia: A total of 3,000 children from Zhongshan Ophthalmic Center is required to undergo ophthalmic examinations and complete questionnaires at baseline and 1yr after wearing Ortho-K.
  Interventions: Device: Orthokeratology lenses

INTERVENTIONS:
Device: Orthokeratology lenses — Orthokeratology lenses

SUMMARY:
This is a prospective study to validate a predictive algorithm for identifying fast progressing myopes.

DETAILED DESCRIPTION:
Orthokeratology (ortho-K) has been demonstrated to slow myopic progression and reduce axial elongation in young patients, but this treatment is limited by the need for contact lens wear, which is the common cause for keratitis in children, and therefore cautious use is recommended. There is a need to identify the patients that could benefit most from this treatment. In order to do so, we conduct a retrospective study and create a large database (n = 10,000) of de-identified data to train an algorithm for identifying fast progressing myopes. In addition, we will perform a prospective study to validate this predictive algorithm and determine the effectiveness of Orthokeratology among different individual patients in China.

ELIGIBILITY:
Inclusion Criteria:

* -6.0D≤SER≤-0.5D
* Astigmatism≤2.0D

Exclusion Criteria:

* Contraindications of wearing Ortho-K.
* Diagnosis of strabismus, amblyopia and other refractive development of the eye or systemic diseases.
* Currently involved in other clinical studies.

Ages: 8 Years to 15 Years | Sex: All
Age Groups: Child
Study Population: 3,000 children from Zhongshan Ophthalmic Center plan to wear orthokeratology lenses for myopia control.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
AUROC of the prediction algorithm for identifying fast progressing myopes | 1 year
  Age-specific axial length (AL) changes previously described by Wang et al.(IOVS, 52 (11), 7949-53, 2011) are used as cut-off values to determine whether a child is a fast progressor or not. A child whose AL change falls on or above the cut-off value is considered to be a fast progressor.

SECONDARY OUTCOMES:
Sensitivity and specificity of the prediction algorithm for identifying fast progressing myopes | 1 year
  The investigators will estimate sensitivity and specificity of the predictive algorithm for identifying fast progressing myopes.
Performance of an algorithm for predicting AL | 1 year
  The investigators will use mean absolute error (MAE), R square to evaluate the performance.
Performance of an algorithm for predicting spherical equivalent refractive error | 1 year
  The investigators will use mean absolute error (MAE), R square to evaluate the performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center (Zhujiang New Town Branch), Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang D, Ding X, Liu B, Zhang J, He M. Longitudinal changes of axial length and height are associated and concomitant in children. Invest Ophthalmol Vis Sci. 2011 Oct 10;52(11):7949-53. doi: 10.1167/iovs.11-7684. PMID 21896861